CLINICAL TRIAL: NCT03687242
Title: A 3-Month Phase 2 Study to Evaluate the Safety and Efficacy of SPR001 in Subjects With Classic Congenital Adrenal Hyperplasia
Brief Title: Study to Evaluate the Safety and Efficacy of SPR001 in Subjects With Classic Congenital Adrenal Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spruce Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR001-202
Record Dates: First submitted 2018-09-11; First posted 2018-09-27 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Congenital Adrenal Hyperplasia; CAH - Congenital Adrenal Hyperplasia; CAH - 21-Hydroxylase Deficiency
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPR001 (Experimental): SPR001 at Dose A
  Interventions: Drug: SPR001

INTERVENTIONS:
Drug: SPR001 — Open label SPR001

SUMMARY:
This is a Phase 2 study of SPR001 for the treatment of classic CAH that will provide 12 weeks of open-label treatment to eligible subjects.

DETAILED DESCRIPTION:
This is a Phase 2 study of SPR001 for the treatment of classic CAH that will provide 12 weeks of open-label treatment to eligible subjects. To be eligible for this study, an individual must either have completed Study SPR001-201 or meet eligibility criteria for SPR001-naïve subjects. The expected duration of study participation for each subject is up to approximately 5 months. This includes a screening period of ≤30 days, a treatment period of 12 weeks, and a safety follow-up period of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Is approved by the Sponsor's Medical Monitor
* Is on a stable regimen of glucocorticoid replacement for ≥30 days before baseline that is expected to remain stable throughout the study
* If screening for this study occurs >3 months after the subject's final follow-up visit in Study SPR001-201, the subject will have serum 17-OHP measured at screening.
* Agrees to follow contraception guidelines
* Is able to understand all study procedures and risks involved and provides written informed consent indicating willingness to comply with all aspects of the protocol

Exclusion Criteria:

* Experienced a clinically significant AE considered at least possibly related to SPR001 in Study SPR001-201
* If screening for this study occurs >3 months after the subject's final follow-up visit in Study SPR001-201, the subject will be screened for any clinically significant unstable medical condition, medically significant illness, or chronic disease occurring within 30 days of screening
* Is at increased risk of suicide
* Clinically significant depression or anxiety at screening or baseline
* Clinically significant abnormal clinical or laboratory assessments must be discussed with the Medical Monitor to determine eligibility for this study.
* Subjects who routinely work overnight shifts require Medical Monitor approval for enrollment
* Females who are pregnant or lactating
* Use of any other investigational drug within 30 days or 5 half-lives before screening
* Use of prohibited concomitant medications (including rosiglitazone, testosterone, and strong inhibitors and/or inducers of CYP3A4) within 30 days or 5 half-lives of baseline. Medications metabolized by CYP3A4, 2C8, 2C9, or 2C19, especially those that are sensitive substrates or substrates with narrow therapeutic ranges should be discussed on a case-by-case basis with the Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Spruce Biosciences
Locations (8):
- United States (8):
  - Spruce Biosciences Clinical Site, Orange, California
  - Spruce Biosciences Clinical Site, San Diego, California
  - Spruce Biosciences Clinical Site, Atlanta, Georgia
  - Spruce Biosciences Clinical Site, Indianapolis, Indiana
  - Spruce Biosciences Clinical Site, Ann Arbor, Michigan
  - Spruce Biosciences Clinical Site, Minneapolis, Minnesota
  - Spruce Biosciences Clinical Site, Las Vegas, Nevada
  - Spruce Biosciences Clinical Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarafoglou K, Barnes CN, Huang M, Imel EA, Madu IJ, Merke DP, Moriarty D, Nakhle S, Newfield RS, Vogiatzi MG, Auchus RJ. Tildacerfont in Adults With Classic Congenital Adrenal Hyperplasia: Results from Two Phase 2 Studies. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4666-e4679. doi: 10.1210/clinem/dgab438. PMID 34146101

RESULTS

PARTICIPANT FLOW:
Groups:
- SPR001: SPR001 at Dose A
  SPR001: Open-label SPR001
Period: Overall Study
Arm/Group | SPR001
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received at least one dose of study drug. This population is the primary analysis set for all efficacy and safety analyses.
Arm/Group | SPR001
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 33.6 (11.31)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Treatment-emergent Adverse Events (Safety and Tolerability) in Subjects With CAH
Description: Incidence of treatment-emergent adverse events including any serious adverse events, dose-limiting toxicities, and adverse events leading to discontinuation of study drug.
Time Frame: Over 12 weeks
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SPR001
Number analyzed (Participants) | 11
Participants
  Subjects experiencing adverse events | 9
  Subjects who did not experience adverse events | 2

2. Secondary Outcome: Change From Baseline in 17-hydroxyprogesterone (17-OHP)
Description: Change from Baseline to Week 12 in 17-OHP following dosing of SPR001 in subjects with CAH. 17-OHP is measured in patient serum sample. Results are expressed as mean percent change from baseline. Reductions in 17-OHP are indicators of better disease control.
Time Frame: Week 12
Population: One subject was withdrawn prematurely on Day 24 due to adverse events and is not included in the efficacy analyses.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | SPR001
Number analyzed (Participants) | 10
percentage of change from baseline | -43.4 (47.83)

3. Secondary Outcome: Change From Baseline in Androstenedione (A4)
Description: Change from Baseline to Week 12 in androstenedione (A4) following dosing of SPR001 in subjects with CAH. A4 is measured in patient serum. Results are expressed as mean percent change from baseline. Reductions in A4 are indicators of better disease control.
Time Frame: Week 12
Population: One subject was withdrawn prematurely on Day 24 due to adverse events and is not included in the efficacy analyses.
Measure: Mean (Standard Deviation); unit: percentage of mean change from baseline
Arm/Group | SPR001
Number analyzed (Participants) | 10
percentage of mean change from baseline | 34.0 (238.20)

4. Secondary Outcome: Change From Baseline in Adrenocorticotropic Hormone (ACTH)
Description: Change from Baseline to Week 12 in adrenocorticotropic hormone (ACTH) following dosing of SPR001 in subjects with CAH. ACTH is measured in patient serum. Results are expressed as mean percent change from baseline. Reductions in ACTH are indicators of better disease control.
Time Frame: Week 12
Population: One subject was withdrawn prematurely on Day 24 due to adverse events and is not included in the efficacy analyses.
Measure: Mean (Standard Deviation); unit: percentage of mean change from baseline
Arm/Group | SPR001
Number analyzed (Participants) | 10
percentage of mean change from baseline | -45.64 (6.244)

ADVERSE EVENTS:
Time Frame: During 12-week treatment period and the 30 days follow-up period, for a total of 16 weeks
Arm/Group | SPR001
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPR001 (N=11)
Hypothyroidism (Endocrine disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03687242/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT03687242/SAP_001.pdf